CLINICAL TRIAL: NCT05030402
Title: Effec of Maitland in Shoulder Pathology
Brief Title: Efficacy of Maitland Mobilization in Shoulder Pathology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Las Palmas de Gran Canaria (Other)
Responsible Party: Principal Investigator, Karishma Chuhermal Lalwani Mangtani, Principal Investigator, University of Las Palmas de Gran Canaria
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ULPGC02
Record Dates: First submitted 2021-06-29; First posted 2021-09-01 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Tendinosis
Keywords: Shoulder; Maitland; Tendinosis
MeSH Terms: conditions — Tendinopathy | interventions — Transcutaneous Electric Nerve Stimulation; Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Maitland group (Experimental): 31 patients receives tens, SW, Maitland, and exercises. An assessment is carried out at the beginning of the treatment, at the end and 2-4 weeks after finishing the treatment. The EVA ASES, DASH and SF-36 scales are included and the biomechanics study is used for the range of mobility.
  Interventions: Procedure: Maitland; Procedure: Tens, exercise, SW
- Control group (Active Comparator): 32 receives tens, SW, conventional physiotherapy and exercises as treatment. An assessment is carried out at the beginning of the treatment, at the end and 2-4 weeks after finishing the treatment. The EVA ASES, DASH and SF-36 scales are included and the biomechanics study is used for the range of mobility.
  Interventions: Procedure: Tens, exercise, SW; Procedure: Conventional physiotherapy

INTERVENTIONS:
Procedure: Maitland — An assessment is carried out at the beginning of the treatment, at the end and 2-4 weeks after finishing the treatment. The EVA ASES, DASH and SF-36 scales are included and the biomechanics study is used for the range of mobility.
  Arms: Maitland group
Procedure: Tens, exercise, SW — An assessment is carried out at the beginning of the treatment, at the end and 2-4 weeks after finishing the treatment. The EVA ASES, DASH and SF-36 scales are included and the biomechanics study is used for the range of mobility.
Procedure: Conventional physiotherapy — An assessment is carried out at the beginning of the treatment, at the end and 2-4 weeks after finishing the treatment. The EVA ASES, DASH and SF-36 scales are included and the biomechanics study is used for the range of mobility.
  Arms: Control group

SUMMARY:
The shoulder is a mobile structure which generates a lot of pathologies. One of them is rotator cuff tendinosis. On the other hand, it has been investigated that Maitland is effective for reducing pain and for mobility in the cervical and lumbar spine and in joints such as the knee and ankle, however, there are few studies that confirm that it is effective in shoulder pathologies.So here the investigatprs want to study the effectiveness of Maitland as an adjunctive treatment for shoulder pathologies, comparing it with conventional physiotherapy treatment, in relation to the reduction of pain and increased mobility. For that the investigators have a randomized clinical trial with two group.

DETAILED DESCRIPTION:
Group 1 receives tens, SW, conventional physiotherapy and exercises as treatment. Group 2 receives tens, SW, Mailtland, and exercises. An assessment is carried out at the beginning of the treatment, at the end and 2-4 weeks after finishing the treatment. The EVA ASES, DASH and SF-36 scales are included and the biomechanics study is used for the range of mobility.

ELIGIBILITY:
Inclusion Criteria:

* Have a shoulder pathology.
* Have a restriction at least of two ranges of movement of the shoulder.
* Sign the consent before starting the study.

Exclusion Criteria:

* Patients with a history of shoulder or neck surgery.
* Patients with neurological damage such as stroke or disease of Parkinson's, as well as those with rheumatism, osteoporosis, surgical fixation, or malignant tumors.
* Have a radiating pain in shoulder from a cervical injury.
* Pregnant patients.
* Patients who do not sign the consent before starting the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2020-09-03 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Change of Range of Motion (ROM) | Baseline and 1, 5, and 7 weeks after treatment
  Active ROM of the affected shoulder is measured using a Mechanic Analysis to assess range of motion. These measurements included abduction, flexion, internal rotation, and external rotation.
Change of Visual Analog Scale (VAS) | Baseline and 1, 5, and 7 weeks after treatment
  Visual analogue score (VAS) was done at rest and at shoulder movement. VAS was explained to the patients during assessment as 0 equal no pain and 10 equal worst imaginable pain.
Change of Disabilities of the Arm, Shoulder and Hand (DASH) | Baseline and 1, 5, and 7 weeks after treatment
  Disabilities of the Arm, Shoulder and Hand (DASH) was filled by patient during assessment as 0 equal better functionality and 100 equal worst functionality

SECONDARY OUTCOMES:
Change of American shoulder and elbow Surgeons" (ASES) | Baseline and 1, 5, and 7 weeks after treatment
  Disabilities of the Arm, Shoulder and Hand (DASH) was filled by patient during assessment as 0 equal worst functionality and 100 is equal better functionality
Change of 36-Item Health Survey (SF-36) | Baseline and 1, 5, and 7 weeks after treatment
  Health Survey (SF-36) was filled by patient during assessment as 0 equal worst health and 100 is equal better health

CONTACTS AND LOCATIONS:
Overall Officials: Karishma LALWANI MANGTAN, Principal Investigator — University of Las Palmas de Gran Canaria (ULPGC)
Locations (1):
- GRUPO ICOT Policlínico Las Palmas., Las Palmas de Gran Canaria, Las Palmas, Spain

REFERENCES:
- [Background] Haider R, Bashir MS, Adeel M, Ijaz MJ, Ayub A. Comparison of conservative exercise therapy with and without Maitland Thoracic Manipulative therapy in patients with subacromial pain: Clinical trial. J Pak Med Assoc. 2018 Mar;68(3):381-387. PMID 29540872
- [Background] Hauswirth J, Ernst MJ, Preusser ML, Meichtry A, Kool J, Crawford RJ. Immediate effects of cervical unilateral anterior-posterior mobilisation on shoulder pain and impairment in post-operative arthroscopy patients. J Back Musculoskelet Rehabil. 2017;30(3):615-623. doi: 10.3233/BMR-160566. PMID 28035910
- [Background] Cook C, Learman K, Houghton S, Showalter C, O'Halloran B. The addition of cervical unilateral posterior-anterior mobilisation in the treatment of patients with shoulder impingement syndrome: a randomised clinical trial. Man Ther. 2014 Feb;19(1):18-24. doi: 10.1016/j.math.2013.05.007. Epub 2013 Jun 20. PMID 23791561
- [Background] Carlson M, Hadlock T. Physical therapist management following rotator cuff repair for a patient with postpolio syndrome. Phys Ther. 2007 Feb;87(2):179-92. doi: 10.2522/ptj.20050200. Epub 2007 Jan 23. PMID 17244697
- [Background] Noten S, Meeus M, Stassijns G, Van Glabbeek F, Verborgt O, Struyf F. Efficacy of Different Types of Mobilization Techniques in Patients With Primary Adhesive Capsulitis of the Shoulder: A Systematic Review. Arch Phys Med Rehabil. 2016 May;97(5):815-25. doi: 10.1016/j.apmr.2015.07.025. Epub 2015 Aug 15. PMID 26284892